CLINICAL TRIAL: NCT07201688
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Trial of Recombinant Human TNK Tissue-Type Plasminogen Activator for Injection (rhTNK-tPA, Mingfule) in Intravenous Thrombolysis for Acute Ischemic Stroke With Extended Time Window (4.5-24 Hours After Onset).
Brief Title: Phase III Clinical Trial of rhTNK-tPA in Treating Acute Ischemic Stroke With Extended Time Window.
Acronym: TRACE-LATE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Mingfule Pharmaceutical (Guangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MK02-003
Record Dates: First submitted 2025-09-22; First posted 2025-10-01 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Eligible subjects were centrally randomized at a 1:1 ratio to receive either rhTNK-Tpa or placebo treatment, with the two groups proceeding simultaneously and without mutual interference.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Receive rhTNK-tPA administration at 0.25mg/kg, with the maximum dose not exceeding 25mg.
  Interventions: Drug: rhTNK-tPA
- Placebo Group (Placebo Comparator): Receive placebo treatment, administration method and dosage same as rhTNK-tPA
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rhTNK-tPA — Each vial should be dissolved in 3mL of sterile water for injection to prepare a drug solution with a concentration of 5.33mg/mL. Calculate the total drug amount based on the participant's actual body weight, measure the required volume of the drug solution, and ensure the maximum dose does not exceed 25mg. Administer as a single bolus intravenous injection, completing the injection within 5-10 seconds.
  Arms: Experimental Group
Drug: Placebo — One vial is dissolved in 3mL of sterile water for injection. Calculate the total drug amount based on the participant's actual body weight, then measure the required volume of the drug solution. Administer as a single bolus intravenous injection, completing the injection within 5-10 seconds.
  Arms: Placebo Group

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase III clinical study designed to evaluate the efficacy of recombinant human tissue-type plasminogen activator variant (rhTNK-tPA) (0.25 mg/kg, maximum dose 25 mg) compared with placebo in patients with acute large vessel occlusive stroke who present within 4.5 to 24 hours of symptom onset. The study plans to enroll patients with acute large vessel occlusive stroke who present within 4.5 to 24 hours of symptom onset (including wake-up strokes and strokes without witnesses). A centralized 1:1 randomization will be adopted, and eligible participants will be randomly assigned to two groups: the experimental group will receive rhTNK-tPA at a dose of 0.25 mg/kg, while the placebo group will receive rhTNK-tPA placebo.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled Phase III clinical study aims to evaluate the efficacy of recombinant human tissue-type plasminogen activator variant (rhTNK-tPA) (0.25 mg/kg, maximum dose 25 mg) compared with placebo in patients with acute large vessel occlusive stroke who present within 4.5 to 24 hours of symptom onset. The study initially planned to enroll 890 patients, who would be randomly assigned to the experimental group (rhTNK-tPA group) or the control group (placebo group) at a 1:1 ratio. After an unblinded sample size re-estimation during the interim analysis, the maximum sample size could be adjusted to 1,300 patients.

Key characteristics of the primary study population include: age ≥ 18 years; time from symptom onset to treatment ranging from 4.5 hours to 24 hours; occlusion of the internal carotid artery, M1 or M2 segment of the middle cerebral artery confirmed by computed tomography angiography (CTA)/magnetic resonance angiography (MRA), which is the responsible vessel for the signs and symptoms of acute ischemic stroke; modified Rankin Scale (mRS) score ≤ 1 before symptom onset; baseline National Institutes of Health Stroke Scale (NIHSS) score ≥ 6; and presence of target mismatch on computed tomography perfusion (CTP) or magnetic resonance imaging (MRI) combined with magnetic resonance perfusion (MRP) (ischemic core volume < 70 mL, mismatch ratio ≥ 1.8, and mismatch volume ≥ 15 mL). Patients with a known allergy to rhTNK-tPA and those with contraindications to thrombolysis were excluded.

The entire study duration is approximately 90 days, including the screening period, treatment period, and follow-up period. The primary study endpoint is the proportion of participants with a modified Rankin Scale (mRS) score of 0-1 at the 90-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years, regardless of gender;
2. Time from symptom onset to treatment is 4.5 - 24 hours(Including the boundary values.), including patients with wake-up stroke or stroke without witnesses; the time of symptom onset is defined as the "last known normal time";
3. Modified Rankin Scale (mRS) score ≤ 1 before stroke onset;
4. Baseline National Institutes of Health Stroke Scale (NIHSS) score ≥ 6;
5. Neuroimaging findings: occlusion of the internal carotid artery (ICA), M1 or M2 segment of the middle cerebral artery (MCA) confirmed by computed tomography angiography (CTA)/magnetic resonance angiography (MRA), which is the responsible vessel for the signs and symptoms of acute ischemic stroke; presence of target mismatch on computed tomography perfusion (CTP) or magnetic resonance imaging (MRI) + magnetic resonance perfusion (MRP) (ischemic core volume < 70 mL, mismatch ratio ≥ 1.8, mismatch volume ≥ 15 mL);
6. Voluntary signing of the informed consent form by the participant or their legal guardian.

Exclusion Criteria:

1. Patients with known allergy to recombinant human tissue plasminogen activator (rhTNK-tPA);
2. Patients with an expected life expectancy of less than 1 year;
3. Patients with rapidly improving symptoms (which may indicate spontaneous recanalization), as determined by the investigator;
4. Patients with a score of > 2 on Item 1a (Level of Consciousness) of the National Institutes of Health Stroke Scale (NIHSS), or those who had a seizure at stroke onset, or had hemiplegia after seizure, or had other neurological/psychiatric disorders that rendered them unable or unwilling to cooperate;
5. Severe and persistent hypertension uncontrolled by medication ;
6. Blood glucose < 2.8 mmol/L or > 22.2 mmol/L;
7. Active internal bleeding with a high risk of hemorrhage;
8. Any known coagulation disorder;
9. Known platelet function defect or platelet count less than 100×10⁹/L;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 890 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with a score of 0-1 on the modified Rankin Scale (mRS) | At Day90.
  The modified Rankin Scale (mRS) is used to assess the status of neurological function recovery in patients after stroke. By evaluating the independence of patients in daily activities, it classifies functional levels into grades 0-6 (Grade 0 indicates no symptoms at all, Grades 1-5 correspond to functional impairments ranging from mild to severe, and Grade 6 indicates death).

SECONDARY OUTCOMES:
Incidence of symptomatic intracerebral hemorrhage within 36 hours after randomization | 36 Hours after Randomization
  Defined by ECASS III: any intraparenchymal or intracranial hemorrhage associated with clinical deterioration, where the latter is defined as an increase of ≥4 points in the National Institutes of Health Stroke Scale [NIHSS] score or death, with confirmation that the hemorrhage is the cause of neurological deterioration.
Overall mortality rate at Day 90. | At Day90.
  The proportion of randomized patients who died within 90 days
Incidence of significant systemic hemorrhage (moderate to severe per GUSTO classification) at Day 90. | At Day90.
  For the Global Use of Strategies to Open Occluded Arteries (GUSTO) Classification, its core lies in categorizing bleeding into three grades-mild, moderate, and severe-based on the impact of bleeding on the patient's clinical status, treatment needs, and prognosis.
Proportion of adverse events (AEs)/serious adverse events (SAEs) at Day 90. | At Day90.
  Adverse Event (AE) refers to any adverse medical event that occurs in a participant after administration of an investigational medicinal product. It may present as signs, symptoms, diseases, or abnormal laboratory findings, but it is not necessarily causally related to the investigational medicinal product. A Serious Adverse Event (SAE) refers to a special safety event among AEs that meets any of the following criteria: "resulting in death, life-threatening, requiring hospitalization/prolongation of existing hospitalization, causing permanent or severe disability/incapacity, leading to congenital anomalies/birth defects, or being another important medical event".
Modified Rankin Scale (mRS) score at Day 90 (shift analysis). | At Day90.
  The modified Rankin Scale (mRS) is used to assess the status of neurological function recovery in patients after stroke. By evaluating the independence of patients in daily activities, it classifies functional levels into grades 0-6 (Grade 0 indicates no symptoms at all, Grades 1-5 correspond to functional impairments ranging from mild to severe, and Grade 6 indicates death).
Title: Proportion of participants with mRS score of 0-2 at Day 90. | At Day90.
  The modified Rankin Scale (mRS) is used to assess the status of neurological function recovery in patients after stroke. By evaluating the independence of patients in daily activities, it classifies functional levels into grades 0-6 (Grade 0 indicates no symptoms at all, Grades 1-5 correspond to functional impairments ranging from mild to severe, and Grade 6 indicates death).
Proportion of participants with an NIHSS score of ≤1 or a reduction of ≥8 points from baseline within 72 hours after randomization. | 72 Hours after Randomization.
  The National Institutes of Health Stroke Scale (NIHSS) is a globally accepted tool for assessing the severity of stroke. Primarily used in patients with acute stroke, it evaluates 11 neurological domains including consciousness, gaze, visual fields, facial palsy, limb motor function, sensation, and language. Scores ranging from 0 to 42 are assigned based on the degree of impairment, where a score of 0 indicates normal neurological function and a score of 42 indicates extremely severe impairment.
Change in NIHSS score from baseline at Day 7. | At Day7.
  The National Institutes of Health Stroke Scale (NIHSS) is a globally accepted tool for assessing the severity of stroke. Primarily used in patients with acute stroke, it evaluates 11 neurological domains including consciousness, gaze, visual fields, facial palsy, limb motor function, sensation, and language. Scores ranging from 0 to 42 are assigned based on the degree of impairment, where a score of 0 indicates normal neurological function and a score of 42 indicates extremely severe impairment.
Proportion of participants with a Barthel Index (BI) score of ≥95 at Day 90. | At Day90.
  The Barthel Index (BI) is a commonly used tool to assess the ability of self-care in daily life for patients with functional impairments (such as those with stroke or spinal cord injury). It mainly evaluates whether patients can independently perform 10 daily activities including eating, dressing, walking, and using the toilet, and assigns a score ranging from 0 to 100 based on their ability level: a score of 100 indicates complete self-care, and the lower the score, the higher the degree of dependence on others.
Rate of favorable reperfusion (90% improvement in Tmax >6s compared with prior status) within 24 hours after randomization. | 24 Hours after Randomization.
  The rate of favorable reperfusion is defined as an improvement of 90% or more in the area with Tmax > 6s (compared with the previous status) on imaging examinations.
Growth of irreversible cerebral infarction volume before treatment and 24 hours after treatment. | 72 Hours after Treatment.
  The volume of irreversible cerebral infarction refers to the brain tissue that has suffered irreversible damage after ischemia, and is also called the volume of core infarction.
Proportion of participants with favorable reperfusion (TICI 2b/3 or TICI 3) on angiography before endovascular treatment (limited to participants who received endovascular treatment). | Periprocedural
  The Thrombolysis in Cerebral Infarction (TICI) Scale is a standard for assessing the degree of cerebral vascular recanalization in patients with acute ischemic stroke after endovascular treatment. It evaluates the blood flow recovery of the infarct-related artery via imaging examinations and is mainly categorized into Grades 0 to 3: Grade 0 represents no perfusion, Grade 1 mild perfusion, Grade 2 partial perfusion, and Grade 3 complete perfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Puyang Oilfield General Hospital, Puyang, Henan, China